CLINICAL TRIAL: NCT03575390
Title: The Beneficial Effects of Pomegranate on Hearing of Patients Without Hemodialysis: A Prospective, Randomized, Double-blinded Clinical Trial
Brief Title: The Beneficial Effects of Pomegranate on Hearing of Patients Without Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dalin Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: B10601002-3
Record Dates: First submitted 2018-01-11; First posted 2018-07-02 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Hearing Impairment
Keywords: Pomegranate; Hearing
MeSH Terms: conditions — Hearing Loss | interventions — maltodextrin; pomegranate fruit rind

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Placebo Comparator): Control group will receive placebo medication therapy
  Interventions: Dietary Supplement: Placebo
- test group (Experimental): pomegranate group will receive oral pomegranate (500 mg, twice per day)
  Interventions: Dietary Supplement: Pomegranate

INTERVENTIONS:
Dietary Supplement: Placebo — The gel contains a mixture of glucose and maltodextrin - a complex carbohydrate - along with fat and a trace of protein.
  Other Names: Maltodextrin
  Arms: control group
Dietary Supplement: Pomegranate — Pomegranate extract 500mg
  Other Names: Pomegranate extract
  Arms: test group

SUMMARY:
Pomegranate has anti-oxidative capacity. It might reduce symptoms of Alzheimer's disease, Drug-induced hepatitis, and might prevent deterioration of cardiovascular diseases and cancer progression. But, the beneficial effects of pomegranate on hearing impairment was still unclear.

This study aimed to investigate the beneficial effects of pomegranate on hearing impairment by a prospective, randomized, double-blinded clinical trial design. The investigators'll include 120 elderly patients without hemodialysis in our hospital, and divided them into 2 groups. Control group will receive placebo treatment; pomegranate group will receive oral pomegranate (500 mg, twice per day).

All patients received the above treatment for 9 months, and underwent pure tone audiometry and word discrimination scores before the start of the clinical trial and at the end of the treatment (9th month).

DETAILED DESCRIPTION:
Pomegranate has anti-oxidative capacity. It might reduce symptoms of Alzheimer's disease, Drug-induced hepatitis, and might prevent deterioration of cardiovascular diseases and cancer progression. But, the beneficial effects of pomegranate on hearing impairment was still unclear.

This study aimed to investigate the beneficial effects of pomegranate on hearing impairment by a prospective, randomized, double-blinded clinical trial design. The investigators'll include 120 elderly patients without hemodialysis in our hospital, and divided them into 2 groups. Control group will receive placebo treatment; pomegranate group will receive oral pomegranate (500 mg, twice per day).

All patients received the above treatment for 9 months, and underwent pure tone audiometry and word discrimination scores before the start of the clinical trial and at the end of the treatment (9th month).

<background> Age-related hearing impairment (ARHI) was very common in the elderly. Hearing deteriorated not only due to problems with the peripheral hearing organs, but also because of degeneration of the central auditory system. In general, peripheral hearing deteriorates more quickly and severely in male subjects than in female subjects, more severely at higher than low frequencies, and more quickly in the central auditory system than the peripheral hearing organs.

1.

Mechanisms of ARHI:

In addition to genetic susceptibility, environmental factors, including obesity, obstructive sleep apnea, systemic diseases, noise, chemical exposure, alcohol, tobacco, ototoxic medication, diet, hormonal factors, menopause and socioeconomic status, may also contribute to hearing degeneration. Contributing mechanisms of this disease may include hypoxia/ischemia, reactive species formation, oxidative stress, and apoptotic/necrotic death of inner ear hair cells/spiral ganglion cells, neural cells, or vascular endothelial cells.

Poor serum vitamin B-12 and folate status levels may be associated with age-related auditory dysfunction in older females. Elevated plasma methylmalonic acid (MMA) concentration may be associated with hearing loss in older adults. Hearing function of noise-exposed workers was negatively correlated with plasma vitamin E levels.

But, one report reported that plasma levels of homocysteine, erythrocyte folate and vitamin B6 were not associated with severity of age-related hearing impairment. Serum magnesium and vitamin C levels were also not correlated with severity of noise-induced hearing loss. The glutathione peroxidase (GPx) 6 gene was upregulated while the thioredoxin reductase 1 gene was downregulated in mice with ARHI. Furthermore, our study group had found that plasma reactive oxygen species levels were correlated with severity of ARHI in humans.

2.

Prevention and/or treatment of ARHI It is reasonable to expect that improved endogenous antioxidant capacity and/or exogenous antioxidant supplementation may suppress oxidative damage to the cells of auditory system.

Some agents were reported to be beneficial for the senescent auditory system. For example, (-)-Epigallocatechin-3-gallate(EGCG) could protect cultured spiral ganglion cells from hydrogen peroxide-induced oxidizing damage. Vitamin C or E could prevent ARHI in animals. Coffee and caffeine were good for auditory neuropathy of mice. Also, antioxidants were also beneficial for the senescent auditory cortex of aged rats. B12 supplementation could prevent hearing loss in B12-deficient individuals. Folic acid supplementation slowed hearing decline slightly in low frequencies, but not in high frequencies in a population without folic acid fortification of food. Higher folate intake had lower risk of developing hearing loss in older males. Coenzyme Q10 (CoQ10) could slow down the deterioration of presbycusis. There was an inverse association between higher intakes of long-chain n23 poly-unsaturated fatty acid (PUFAs) and regular weekly consumption of fish and age-related hearing loss. Patients who achieved the highest plasma concentrations of vitamin C, vitamin E and selenium had significantly less loss of high-tone hearing. And, salicylate use and moderate alcohol intake were possible protective factors for ARHI.

But, report claimed that life style with higher intake of vitamin C, E, beta carotene, or B12 did not reduce the risk of hearing loss in adult males. Vitamin E or atorvastatin cannot slow down the deterioration of presbycusis. Low-dose difluoromethylornithine (DFMO) could not protect hearing.

3.

Introduction of pomegranate:

Pomegranate is a subtropical and tropical fruit of great importance from a health point of view. It has antioxidant activity and antimutagenic potential. Oxidative and histologic evaluation showed that pomegranate juice might have a preventive effect in paracetamol-induced acute liver damage. Six weeks supplementation of pomegranate juice could have favorable effects on oxidative stress in patients with type 2 diabetes. Pomegranate extract alleviates disease activity and some blood biomarkers of inflammation and oxidative stress in rheumatoid arthritis patients.

Pomegranate seed extract exhibited therapeutic potential for memory and muscular coordination in rats, which was most likely related at least in some part to its antioxidative and free radical scavenging actions. Long-term dietary supplementation with pomegranates from Oman attenuates cognitive and behavioral deficits in a transgenic mice model of Alzheimer's disease. Consumption of pomegranates improves synaptic function in a transgenic mice model of Alzheimer's disease. Pomegranate's neuroprotective effects against Alzheimer's disease are mediated by urolithin, its ellagitannin-gut microbial derived metabolites.

A systematic review and meta-analysis of randomized controlled trials (RCTs) did not suggest any effect of pomegranate consumption on lipid profile and on plasma c-reactive protein levels. One report also concluded that the quality of previous studies about the use of dietary pomegranate preparations in the prevention and treatment of cardiovascular diseases was poor. Even in the best studies, indications of benefit did not reach the conventional levels of statistical significance. And, future studies need to prove the clinical benefit.

Methanol extract of pericarp of pomegranate (PME) had anti-proliferative effect on human breast (MCF-7, MDA-MB-231), endometrial (HEC-1A), cervical (SiHa, HeLa), and ovarian (SKOV3) cancer cell lines, and normal breast fibroblasts (MCF-10A). Also, PME could modulate osteoblastic cell differentiation. Pomegranate evokes antiproliferative, anti-invasive, and antimetastatic effects, induces apoptosis through the modulation of Bcl-2 proteins, upregulates p21 and p27, and downregulates cyclin-cdk network. Furthermore, pomegranate blocks the activation of inflammatory pathways including, but not limited to, the nuclear factor kappa-light-chain-enhancer of activated B cells(NF-κB) pathway. However, another meta-analysis showed that the evidence of clinical effectiveness for cancer treatment in humans was poor because the quality of the studies was poor.

4.

Pomegranate:

A new candidate for ARHI treatment? Pomegranate has antioxidative capacity and could prevent Alzheimer's disease. Meanwhile, oxidative damage was one of the underlying mechanisms for ARHI. So, it is reasonable to expect that pomegranate might have a beneficial effect for ARHI.

ELIGIBILITY:
Inclusion Criteria:

1. Age 50 to 80 years old.
2. non-renal dialysis patients.

Exclusion Criteria:

1. Life can not take care of themselves or the bed of a patient.
2. dialysis patients.
3. Patients who can not understand the details of this study or are unable to cooperate with the examination.
4. history of alcohol or drug abuse.
5. history of high environmental noise exposure.
6. The pure tone hearing threshold is greater than 10 decibel (dB), and the audiogram 4 kilohertz (kHz) air conduction threshold is greater than 8 kilohertz (kHz) air threshold value of 20 decibel (dB).

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-03-30 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Pure tone audiometry (PTA) | 9 months
  pure tone thresholds of 250, 500, 1000, 2000, 4000, 8000 Hz were measured.

SECONDARY OUTCOMES:
speech reception threshold (SRT) | 9 months
  The speech recognition threshold is the lowest hearing level at which speech can barely be recognized or understood. The SRT is defined as the lowest hearing level at which the patient correctly repeats 50% of a list of spondaic words. Examples are airplane, hot dog, outside, ice cream, and baseball. Usually a very soft level (db HL).
speech discrimination score (SDS) | 9 months
  The SDS test tool is a single syllable word list. Each table consists of 50 words, such as, look, go. The test method is to listen to the subject at a volume higher than the SRT value of 20 to 40 dB (30 dB), so that the subject repeats the spoken word sound. Based on the percentage of correct answers, normal people can repeat 95 to 100% of the words, and 80% or less of them are bad discriminating power and affect the understanding of language. SDS is usually expressed in %.

CONTACTS AND LOCATIONS:
Overall Officials: Juen-Haur Hwang, MD, PhD., Study Chair — Dalin Tzu Chi Hospital
Locations (1):
- Dalin Tzu Chi Hospital, Chiayi City, Taiwan